CLINICAL TRIAL: NCT03687567
Title: A Retrospective Study on the Effect of HBA or HBB Genetic Defects on Early Embryonic Development
Status: Completed | Type: Observational
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Other Study IDs: KYXM-201804
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Thalassemia,Embryonic Development,Reproductive Sterility and Infertility
MeSH Terms: conditions — Thalassemia; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBA: alpha-Thalassemia
  Interventions: Procedure: Preimplantation genetic diagnosis
- HBB: beta-Thalassemia
  Interventions: Procedure: Preimplantation genetic diagnosis

INTERVENTIONS:
Procedure: Preimplantation genetic diagnosis

SUMMARY:
Thalassemia is an anemia or pathological state caused by compounding absently or inadequately of one or more globin chains of hemoglobin due to the defects of the globin gene,and the carrying rate is high in southern China. Although there are many studies of Thalassemia, the relationship between the globin gene defects and the early embryo development has not been reported.

This study intends to carry out a retrospective analysis on the embryonic development of the patients with thalassemia assisted by PGD from January 1, 2011 to now in our hospital, to explore whether the HBA or HBB gene defects have a certain influence on the early embryo development, so as to accumulate certain data for reproductive health research.

ELIGIBILITY:
Inclusion Criteria:

* infertility couples with thalassemia(one or both )
* infertility couples treat by PGD

Exclusion Criteria:

* abortion of amplification for blastula biopsy
* PGD without diagnostic results or with unclear diagnostic results
* embryos with both HBA and HBB genetic defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One or both of infertility couples with thalassemia take PGD treatment.
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Gardner grading of blastocysts | embryo cultured in-vitro for 5-7 days
  development status of blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Liang Hu, MD,PHD, Principal Investigator — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided